CLINICAL TRIAL: NCT06024330
Title: External Validation of the VAN, VES, and LARIO Scoring Systems in Patients Suspected of Acute Stroke in Emergency Triage: A Multicenter Prospective Cross-sectional Study
Brief Title: External Validation of VAN, VES and LARIO Scales in Suspected Acute Stroke
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Ibrahim Ulas Ozturan, Assistant Professor, Kocaeli University
Other Study IDs: KU GOEK-2022/06.15
Record Dates: First submitted 2023-08-29; First posted 2023-09-06 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: Triage; Emergency Departments; Stroke; Scales
MeSH Terms: conditions — Stroke; Emergencies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Positive VAN scale: Motor Function: Check for arm drift with arms extended, palms up, and eyes closed for 10 seconds. If present, proceed to the VAN criteria.
  V (Visual): Assess for reported double vision, field cut, or vision loss, or difficulty seeing fingers in a quadrant. If any visual disturbances are found, the patient is "VAN positive".
  A (Aphasia): Identify difficulties forming words, repeating a short sentence, recognizing two objects, or following simple commands. If any aphasia symptoms are observed, the patient is "VAN positive".
  N (Neglect): Check for forced gaze, inability to track a pen to one side, or lack of sensation in limbs. If any neglect signs are detected, the patient is "VAN positive".
  Interventions: Diagnostic Test: VAN assessment
- Negative VAN scale: A negative VAN scale indicates that a potential stroke patient does not exhibit the primary signs associated with a large vessel occlusion (LVO). Specifically, the patient demonstrated no arm drift during the initial motor function test. If the motor assessment is proceeded to the VAN criteria, the patient shows no visual disturbances like double vision or field cuts ("V"), no aphasia symptoms such as difficulty forming words or repeating sentences ("A"), and no signs of neglect, like forced gaze or lack of sensation in limbs ("N")
  Interventions: Diagnostic Test: VAN assessment
- Positive VES scale: Eye Deviation: Scored as 1 if there's a forced deviation of both eyes to any side; otherwise, scored as 0.
  Aphasia: Scored as 1 if the patient is awake and exhibits one or more of the following:
  Inability to repeat a sentence. Inability to name an object. Talking incoherently or not obeying commands. Being mute. Otherwise, scored as 0. Neglect: Scored as 1 if the patient can perceive touch on both sides individually but fails to feel it on one side when stimulated simultaneously. Otherwise, scored as 0.
  Obtundation: Scored as 1 if the patient cannot maintain wakefulness during a conversation; otherwise, scored as 0.
  The VES can range from 0 to 4. A score of 1 or higher suggests a positive likelihood for ELVO. Additionally, if a patient tests positive for aphasia, neglect can be deduced by noting if the patient disregards the examiner on one side but is responsive when the examiner switches sides.
  Interventions: Diagnostic Test: VES assessment
- Negative VES scale: Eye Deviation: No forced deviation of both eyes is observed. Aphasia: The patient, while awake, can repeat sentences, name objects, speaks coherently, follows commands, and is not mute.
  Neglect: The patient can perceive touch both when sides are stimulated individually and simultaneously.
  Obtundation: The patient remains awake and alert during conversation. A total score of 0 on the VES scale represents a VES negative outcome.
  Interventions: Diagnostic Test: VES assessment
- Positive LARIO scale: Facial Palsy: The presence of facial muscle weakness or paralysis scores 1, while a normal facial expression scores 0.
  Arm Weakness: A score of 1 is given for arm drift, no effort against gravity, or no movement at all. No drift is scored 0.
  Grip Strength: Reduced or absent grip strength scores 1, while a normal grip scores 0.
  Language: Changes in speech, global aphasia, or the patient being mute results in a score of 1. Normal language is scored 0.
  Neglect: A score of 1 is given if the patient exhibits extinction to bilateral simultaneous stimulation in one or more sensory modality, doesn't recognize their own hand, or consistently orients only to one side of the body. The absence of these signs scores 0.
  A cumulative score exceeding 3 on the LARIO Stroke Scale categorizes the patient as "LARIO positive,"
  Interventions: Diagnostic Test: LARIO assessment
- Negative LARIO scale: Facial Palsy: No observable facial muscle weakness or paralysis. Arm Weakness: The arm remains steady without drift and exhibits normal effort against gravity.
  Grip Strength: The patient displays normal grip strength. Language: The patient speaks normally, without aphasia or muteness. Neglect: No signs of sensory extinction upon bilateral simultaneous stimulation, proper recognition of their own hand, and balanced orientation to both sides of the body.
  A cumulative score of 3 or less on the LARIO Stroke Scale classifies the patient as "LARIO negative,"
  Interventions: Diagnostic Test: LARIO assessment

INTERVENTIONS:
Diagnostic Test: VAN assessment — An investigator assesses the VAN scale when a patient arrives at ED triage with a suspected stroke.
  Groups: Negative VAN scale; Positive VAN scale
Diagnostic Test: VES assessment — An investigator assesses the VES scale when a patient arrives at ED triage with a suspected stroke.
  Groups: Negative VES scale; Positive VES scale
Diagnostic Test: LARIO assessment — An investigator assesses the LARIO scale when a patient arrives at ED triage with a suspected stroke.
  Groups: Negative LARIO scale; Positive LARIO scale

SUMMARY:
In acute ischemic stroke, treatments include intravenous thrombolysis (IVT) and mechanical thrombectomy (MT). IVT is viable up to 4.5 hours post-stroke onset, while MT is applicable within 24 hours but primarily for large vessel occlusions. MT is specialized and performed in select stroke centers. Effective early triage improves neurological outcomes. Pre-hospital stroke severity assessment and direct transfers for MT are crucial. Although the National Institute of Health Stroke Scale (NIHSS) is widely recognized, its practicality is limited in emergency settings due to its complexity. Alternative scoring systems like LAMS, CPSS, and RACE have been introduced but have limitations. Recently developed scores, namely Vision, Aphasia, and Neglect (VAN), Ventura Emergency Large Vessel Occlusion (VES), and Large Artery Intracranial Occlusion Stroke Scale (LARIO), demonstrate promising diagnostic accuracy in pilot studies, suggesting potential benefits for early detection, appropriate triage, and better neurological outcomes

DETAILED DESCRIPTION:
For acute ischemic stroke, time-dependent treatments include intravenous thrombolysis (IVT) and mechanical thrombectomy (MT). IVT can be considered in all patients with acute ischemic stroke within the first 4.5 hours after the last known well time. However, MT can only be applied within the first 24 hours in large vessel occlusions defined as acute occlusion of the intracranial internal carotid artery (ICA), proximal posterior, middle, and anterior cerebral arteries (respectively PCA, MCA, ACA), intracranial vertebral artery and/or basilar artery. However, MT can only be performed in stroke centers specialized in this area. Effective triage of large vessel occlusion and early application of emergency stroke protocols are associated with good neurological outcomes. In this sense, pre-hospital determination of stroke severity and direct transfer of patients requiring MT to the stroke center are recommended by current guidelines. It is important that the protocols used in pre-hospital and emergency department triage to determine stroke severity are easy to learn and apply, are repeatable, and their accuracy is proven with external data sets. To date, many scoring systems have been proposed for early determination of stroke severity. Although the most accepted and widely used system among these systems is the National Institute of Health Stroke Scale (NIHSS), the need for training and experience for practitioners and the time-consuming application restrict its use in pre-hospital or emergency department triage. Alternatively, short and easily applicable systems such as The Los Angeles Motor Scale (LAMS), The Cincinnati Prehospital Stroke Scale (CPSS), Rapid Arterial oCclusion Evaluation (RACE) have been developed in the pre-hospital setting. However, the inability of these systems to provide high sensitivity and specificity together has necessitated the development of other alternative scoring systems. Among the new scoring systems developed in recent years, the Vision, Aphasia, and Neglect (VAN) score, the Ventura Emergency Large Vessel Occlusion (VES) score, and the Large Artery Intracranial Occlusion Stroke Scale (LARIO) have shown high diagnostic performance in pilot studies. The VAN score was shown to be 100% sensitive and 90% specific in predicting large vessel occlusion in stroke patients with motor weakness accompanied by at least one of the symptoms of vision, aphasia, and neglect or an NIHSS score of >6. The VES score was developed as a 4-step system evaluating eye deviation, aphasia, neglect, and lethargy, and it was reported that the presence of at least one of these functions was 95% sensitive and 82% specific in predicting large vessel occlusion. The LARIO score was developed as a 5-step system evaluating facial paralysis, speech disorder, arm weakness, hand grip weakness, and neglect. Having >3 of these steps positive provided 100% sensitivity and 82% specificity for large vessel occlusion. The results obtained from pilot studies suggest that the use of VAN, VES, and LARIO scoring systems in pre-hospital or emergency department triage promises to improve neurological outcomes by early identification of patients with large vessel occlusion requiring MT, appropriate triage, and optimal application of stroke protocols

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the ED with the suspicion of stroke by EMS.

Exclusion Criteria:

* More than 24 hours have passed since the onset of symptoms or the last known normal in the patient.
* The emergency physician does not indicate the need for imaging like Computerized Tomography (CT), CT Angiography (CTA), Diffusion-Weighted Magnetic Resonance Imaging (DWI-MRI), or Magnetic Resonance Angiography (MRA), or the imaging test cannot be performed.
* Exacerbation of residual symptoms due to a previous hemorrhagic or ischemic stroke.
* Conditions in the ED that prevent scale assessment (e.g., advanced airway needs, the patient's non-cooperation with the examination, immediate resuscitation need, etc.).
* Patients transferred to ED after being diagnosed at another healthcare institution.
* Pregnant patients
* Non-consenting patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All eligible patients with a suspicion of stroke who were admitted to the ED by EMS.
Sampling Method: Non-Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of VAN for predicting ELVO | 24 hours
  Sensitivity, specificity, PPV, NPV
Diagnostic performance of VES for predicting ELVO | 24 hours
  Sensitivity, specificity, PPV, NPV
Diagnostic performance of LARIO for predicting ELVO | 24 hours
  Sensitivity, specificity, PPV, NPV

SECONDARY OUTCOMES:
Diagnostic performance of NIHSS for predicting ELVO | 24 hours
  Sensitivity, specificity, PPV, NPV

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, İzmit, Kocaeli, Turkey (Türkiye)